CLINICAL TRIAL: NCT06854107
Title: Intratumoral and Peritumoral Habitat Radiomics of MRI Predict Pathologic Complete Response to Neoadjuvant Chemoimmunotherapy in Oral Squamous Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Zilong Yuan (Other)
Collaborators: Hubei Cancer Hospital (Other)
Responsible Party: Sponsor-Investigator, Zilong Yuan, Clinical Professor, Hubei Cancer Hospital
Organization: Hubei Cancer Hospital (Other)
Other Study IDs: [2024]KYLL(SO4); no. 2025HBCHHHRC006 (Other Grant/Funding Number: Yuan Wu)
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Pathologic Complete Response
Keywords: Oral squamous cell carcinoma; Radiomics; Intratumoral and peritumoral; Habitat imaging; Pathologic complete response
MeSH Terms: conditions — Pathologic Complete Response; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background：Neoadjuvant chemoimmunotherapy (NACI) shows promise in oral squamous cell carcinoma (OSCC), but reliable noninvasive biomarkers for predicting pathologic complete response (pCR) remain scarce. Radiomics integrating intratumoral and peritumoral heterogeneity across multi-sequence MRI may offer novel insights into treatment response evaluation.

Methods: The data of 212 patients with OSCC after NACI were retrospectively collected and analyzed. Among these patients, 56 (26.4%) achieved pCR after NACI. Intratumoral and peritumoral habitat imaging (HI) was achieved using the K-means clustering algorithm applied to T1-weighted imaging (T1WI), axial T2-weighted imaging with fat suppression (T2WI), and contrast-enhanced T1-weighted imaging with fat suppression (T1C). Moreover, intratumoral and peritumoral HI models were constructed and compared using the receiver operating characteristic (ROC) curve. Five-fold cross-validation was performed to mitigate model overfitting.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed OSCC at the initial diagnosis;
* No treatment received prior to the first MRI examination;
* Receipt of NACI;
* Underwent MRI examination after NACI;
* Underwent surgical intervention.

Exclusion Criteria:

* Absence of clinical data and postoperative pathological results;
* MRI image artifacts significantly affecting image quality.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study comprehensively reviewed the clinical information of OSCC patients who underwent NACI at two institutions from March 2020 to December 2023.
Sampling Method: Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Intratumoral and Peritumoral Habitat Radiomics of MRI predicts pathologic complete response to neoadjuvant chemoimmunotherapy in oral squamous cell carcinoma | From 2024 to 2025
  Integrated intratumoral and peritumoral HI derived from multi-sequence MRI offers a high predictive capacity for pCR following NACI in OSCC patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Hubei Cancer Hospitla, Wuhan, Hubei, China

REFERENCES:
- [Background] Vaidya P, Bera K, Patil PD, Gupta A, Jain P, Alilou M, Khorrami M, Velcheti V, Madabhushi A. Novel, non-invasive imaging approach to identify patients with advanced non-small cell lung cancer at risk of hyperprogressive disease with immune checkpoint blockade. J Immunother Cancer. 2020 Oct;8(2):e001343. doi: 10.1136/jitc-2020-001343. PMID 33051342
- [Background] Tunali I, Hall LO, Napel S, Cherezov D, Guvenis A, Gillies RJ, Schabath MB. Stability and reproducibility of computed tomography radiomic features extracted from peritumoral regions of lung cancer lesions. Med Phys. 2019 Nov;46(11):5075-5085. doi: 10.1002/mp.13808. Epub 2019 Sep 23. PMID 31494946
- [Background] Wang CY, Ginat DT. Preliminary Computed Tomography Radiomics Model for Predicting Pretreatment CD8+ T-Cell Infiltration Status for Primary Head and Neck Squamous Cell Carcinoma. J Comput Assist Tomogr. 2021 Jul-Aug 01;45(4):629-636. doi: 10.1097/RCT.0000000000001149. PMID 34519454
- [Background] Wang C, Wu F, Wang F, Chong HH, Sun H, Huang P, Xiao Y, Yang C, Zeng M. The Association Between Tumor Radiomic Analysis and Peritumor Habitat-Derived Radiomic Analysis on Gadoxetate Disodium-Enhanced MRI With Microvascular Invasion in Hepatocellular Carcinoma. J Magn Reson Imaging. 2025 Mar;61(3):1428-1439. doi: 10.1002/jmri.29523. Epub 2024 Jul 12. PMID 38997242
- [Background] Shang Y, Chen W, Li G, Huang Y, Wang Y, Kui X, Li M, Zheng H, Zhao W, Liu J. Computed Tomography-derived intratumoral and peritumoral radiomics in predicting EGFR mutation in lung adenocarcinoma. Radiol Med. 2023 Dec;128(12):1483-1496. doi: 10.1007/s11547-023-01722-6. Epub 2023 Sep 25. PMID 37749461
- [Background] Shang Y, Zeng Y, Luo S, Wang Y, Yao J, Li M, Li X, Kui X, Wu H, Fan K, Li ZC, Zheng H, Li G, Liu J, Zhao W. Habitat Imaging With Tumoral and Peritumoral Radiomics for Prediction of Lung Adenocarcinoma Invasiveness on Preoperative Chest CT: A Multicenter Study. AJR Am J Roentgenol. 2024 Oct;223(4):e2431675. doi: 10.2214/AJR.24.31675. Epub 2024 Aug 14. PMID 39140631
- [Background] Jiang Y, Wang H, Wu J, Chen C, Yuan Q, Huang W, Li T, Xi S, Hu Y, Zhou Z, Xu Y, Li G, Li R. Noninvasive imaging evaluation of tumor immune microenvironment to predict outcomes in gastric cancer. Ann Oncol. 2020 Jun;31(6):760-768. doi: 10.1016/j.annonc.2020.03.295. Epub 2020 Mar 30. PMID 32240794
- [Background] Braman N, Prasanna P, Whitney J, Singh S, Beig N, Etesami M, Bates DDB, Gallagher K, Bloch BN, Vulchi M, Turk P, Bera K, Abraham J, Sikov WM, Somlo G, Harris LN, Gilmore H, Plecha D, Varadan V, Madabhushi A. Association of Peritumoral Radiomics With Tumor Biology and Pathologic Response to Preoperative Targeted Therapy for HER2 (ERBB2)-Positive Breast Cancer. JAMA Netw Open. 2019 Apr 5;2(4):e192561. doi: 10.1001/jamanetworkopen.2019.2561. PMID 31002322
- [Background] Wu J, Cao G, Sun X, Lee J, Rubin DL, Napel S, Kurian AW, Daniel BL, Li R. Intratumoral Spatial Heterogeneity at Perfusion MR Imaging Predicts Recurrence-free Survival in Locally Advanced Breast Cancer Treated with Neoadjuvant Chemotherapy. Radiology. 2018 Jul;288(1):26-35. doi: 10.1148/radiol.2018172462. Epub 2018 May 1. PMID 29714680
- [Background] Xie C, Yang P, Zhang X, Xu L, Wang X, Li X, Zhang L, Xie R, Yang L, Jing Z, Zhang H, Ding L, Kuang Y, Niu T, Wu S. Sub-region based radiomics analysis for survival prediction in oesophageal tumours treated by definitive concurrent chemoradiotherapy. EBioMedicine. 2019 Jun;44:289-297. doi: 10.1016/j.ebiom.2019.05.023. Epub 2019 May 23. PMID 31129097
- [Background] Wu J, Gensheimer MF, Zhang N, Guo M, Liang R, Zhang C, Fischbein N, Pollom EL, Beadle B, Le QT, Li R. Tumor Subregion Evolution-Based Imaging Features to Assess Early Response and Predict Prognosis in Oropharyngeal Cancer. J Nucl Med. 2020 Mar;61(3):327-336. doi: 10.2967/jnumed.119.230037. Epub 2019 Aug 16. PMID 31420498
- [Background] Kim M, Park JE, Yoon SK, Kim N, Kim YH, Kim JH, Kim HS. Vessel size and perfusion-derived vascular habitat refines prediction of treatment failure to bevacizumab in recurrent glioblastomas: validation in a prospective cohort. Eur Radiol. 2023 Jun;33(6):4475-4485. doi: 10.1007/s00330-022-09164-w. Epub 2022 Oct 15. PMID 36242633
- [Background] Lee DH, Park JE, Kim N, Park SY, Kim YH, Cho YH, Kim JH, Kim HS. Tumor Habitat Analysis Using Longitudinal Physiological MRI to Predict Tumor Recurrence After Stereotactic Radiosurgery for Brain Metastasis. Korean J Radiol. 2023 Mar;24(3):235-246. doi: 10.3348/kjr.2022.0492. Epub 2023 Feb 6. PMID 36788768
- [Background] Ling X, Alexander GS, Molitoris J, Choi J, Schumaker L, Mehra R, Gaykalova DA, Ren L. Identification of CT-based non-invasive radiomic biomarkers for overall survival prediction in oral cavity squamous cell carcinoma. Sci Rep. 2023 Dec 8;13(1):21774. doi: 10.1038/s41598-023-48048-x. PMID 38066047
- [Background] Ozturk EMA, Unsal G, Erisir F, Orhan K. Prediction of bone invasion of oral squamous cell carcinoma using a magnetic resonance imaging-based machine learning model. Eur Arch Otorhinolaryngol. 2024 Dec;281(12):6585-6597. doi: 10.1007/s00405-024-08862-z. Epub 2024 Jul 31. PMID 39083062
- [Background] Ling X, Alexander GS, Molitoris J, Choi J, Schumaker L, Tran P, Mehra R, Gaykalova D, Ren L. Radiomic biomarkers of locoregional recurrence: prognostic insights from oral cavity squamous cell carcinoma preoperative CT scans. Front Oncol. 2024 Apr 23;14:1380599. doi: 10.3389/fonc.2024.1380599. eCollection 2024. PMID 38715772
- [Background] Hinzpeter R, Mirshahvalad SA, Kulanthaivelu R, Ortega C, Metser U, Liu ZA, Elimova E, Wong RKS, Yeung J, Jang RW, Veit-Haibach P. Prognostic Value of [18F]-FDG PET/CT Radiomics Combined with Sarcopenia Status among Patients with Advanced Gastroesophageal Cancer. Cancers (Basel). 2022 Oct 28;14(21):5314. doi: 10.3390/cancers14215314. PMID 36358733
- [Background] Tomita H, Yamashiro T, Heianna J, Nakasone T, Kimura Y, Mimura H, Murayama S. Nodal-based radiomics analysis for identifying cervical lymph node metastasis at levels I and II in patients with oral squamous cell carcinoma using contrast-enhanced computed tomography. Eur Radiol. 2021 Oct;31(10):7440-7449. doi: 10.1007/s00330-021-07758-4. Epub 2021 Mar 31. PMID 33787970
- [Background] Jin N, Qiao B, Zhao M, Li L, Zhu L, Zang X, Gu B, Zhang H. Predicting cervical lymph node metastasis in OSCC based on computed tomography imaging genomics. Cancer Med. 2023 Sep;12(18):19260-19271. doi: 10.1002/cam4.6474. Epub 2023 Aug 27. PMID 37635388
- [Background] Chen Z, Yu Y, Liu S, Du W, Hu L, Wang C, Li J, Liu J, Zhang W, Peng X. A deep learning and radiomics fusion model based on contrast-enhanced computer tomography improves preoperative identification of cervical lymph node metastasis of oral squamous cell carcinoma. Clin Oral Investig. 2023 Dec 27;28(1):39. doi: 10.1007/s00784-023-05423-2. PMID 38151672
- [Background] Li W, Li Y, Gao S, Huang N, Kojima I, Kusama T, Ou Y, Iikubo M, Niu X. Integrating lipid metabolite analysis with MRI-based transformer and radiomics for early and late stage prediction of oral squamous cell carcinoma. BMC Cancer. 2024 Jul 3;24(1):795. doi: 10.1186/s12885-024-12533-x. PMID 38961418
- [Background] Liu H, Zhu C, Wang X, Chen X, Li Z, Xian J. Prediction of pathological complete response in locally advanced head and neck squamous cell carcinoma treated with neoadjuvant chemo-immunotherapy using volumetric multisequence MRI histogram analysis. Neuroradiology. 2024 Jun;66(6):919-929. doi: 10.1007/s00234-024-03339-6. Epub 2024 Mar 20. PMID 38503986
- [Background] Yuan Y, Ren J, Shi Y, Tao X. MRI-based radiomic signature as predictive marker for patients with head and neck squamous cell carcinoma. Eur J Radiol. 2019 Aug;117:193-198. doi: 10.1016/j.ejrad.2019.06.019. Epub 2019 Jun 25. PMID 31307647
- [Background] Lin P, Xie W, Li Y, Zhang C, Wu H, Wan H, Gao M, Liang F, Han P, Chen R, Cheng G, Liu X, Fan S, Huang X. Intratumoral and peritumoral radiomics of MRIs predicts pathologic complete response to neoadjuvant chemoimmunotherapy in patients with head and neck squamous cell carcinoma. J Immunother Cancer. 2024 Nov 5;12(11):e009616. doi: 10.1136/jitc-2024-009616. PMID 39500529
- [Background] Yoon H, Ha S, Kwon SJ, Park SY, Kim J, O JH, Yoo IR. Prognostic value of tumor metabolic imaging phenotype by FDG PET radiomics in HNSCC. Ann Nucl Med. 2021 Mar;35(3):370-377. doi: 10.1007/s12149-021-01586-8. Epub 2021 Feb 8. PMID 33554314
- [Background] Alfieri S, Romano R, Bologna M, Calareso G, Corino V, Mirabile A, Ferri A, Bellanti L, Poli T, Marcantoni A, Grosso E, Tarsitano A, Battaglia S, Blengio F, De Martino I, Valerini S, Vecchio S, Richetti A, Deantonio L, Martucci F, Grammatica A, Ravanelli M, Ibrahim T, Caruso D, Locati LD, Orlandi E, Bossi P, Mainardi L, Licitra LF. Prognostic role of pre-treatment magnetic resonance imaging (MRI)-based radiomic analysis in effectively cured head and neck squamous cell carcinoma (HNSCC) patients. Acta Oncol. 2021 Sep;60(9):1192-1200. doi: 10.1080/0284186X.2021.1924401. Epub 2021 May 26. PMID 34038324
- [Background] Ou D, Blanchard P, Rosellini S, Levy A, Nguyen F, Leijenaar RTH, Garberis I, Gorphe P, Bidault F, Ferte C, Robert C, Casiraghi O, Scoazec JY, Lambin P, Temam S, Deutsch E, Tao Y. Predictive and prognostic value of CT based radiomics signature in locally advanced head and neck cancers patients treated with concurrent chemoradiotherapy or bioradiotherapy and its added value to Human Papillomavirus status. Oral Oncol. 2017 Aug;71:150-155. doi: 10.1016/j.oraloncology.2017.06.015. Epub 2017 Jun 26. PMID 28688683
- [Background] Leger S, Zwanenburg A, Leger K, Lohaus F, Linge A, Schreiber A, Kalinauskaite G, Tinhofer I, Guberina N, Guberina M, Balermpas P, von der Grun J, Ganswindt U, Belka C, Peeken JC, Combs SE, Boeke S, Zips D, Richter C, Krause M, Baumann M, Troost EGC, Lock S. Comprehensive Analysis of Tumour Sub-Volumes for Radiomic Risk Modelling in Locally Advanced HNSCC. Cancers (Basel). 2020 Oct 19;12(10):3047. doi: 10.3390/cancers12103047. PMID 33086761
- [Background] Mes SW, van Velden FHP, Peltenburg B, Peeters CFW, Te Beest DE, van de Wiel MA, Mekke J, Mulder DC, Martens RM, Castelijns JA, Pameijer FA, de Bree R, Boellaard R, Leemans CR, Brakenhoff RH, de Graaf P. Outcome prediction of head and neck squamous cell carcinoma by MRI radiomic signatures. Eur Radiol. 2020 Nov;30(11):6311-6321. doi: 10.1007/s00330-020-06962-y. Epub 2020 Jun 4. PMID 32500196
- [Background] Keek S, Sanduleanu S, Wesseling F, de Roest R, van den Brekel M, van der Heijden M, Vens C, Giuseppina C, Licitra L, Scheckenbach K, Vergeer M, Leemans CR, Brakenhoff RH, Nauta I, Cavalieri S, Woodruff HC, Poli T, Leijenaar R, Hoebers F, Lambin P. Computed tomography-derived radiomic signature of head and neck squamous cell carcinoma (peri)tumoral tissue for the prediction of locoregional recurrence and distant metastasis after concurrent chemo-radiotherapy. PLoS One. 2020 May 22;15(5):e0232639. doi: 10.1371/journal.pone.0232639. eCollection 2020. PMID 32442178
- [Background] Wang K, Zhou Z, Wang R, Chen L, Zhang Q, Sher D, Wang J. A multi-objective radiomics model for the prediction of locoregional recurrence in head and neck squamous cell cancer. Med Phys. 2020 Oct;47(10):5392-5400. doi: 10.1002/mp.14388. Epub 2020 Aug 5. PMID 32657426
- [Background] Katsoulakis E, Yu Y, Apte AP, Leeman JE, Katabi N, Morris L, Deasy JO, Chan TA, Lee NY, Riaz N, Hatzoglou V, Oh JH. Radiomic analysis identifies tumor subtypes associated with distinct molecular and microenvironmental factors in head and neck squamous cell carcinoma. Oral Oncol. 2020 Nov;110:104877. doi: 10.1016/j.oraloncology.2020.104877. Epub 2020 Jun 30. PMID 32619927
- [Background] Wu D, Li Y, Xu P, Fang Q, Cao F, Lin H, Li Y, Su Y, Lu L, Chen L, Li Y, Zhao Z, Hong X, Li G, Tian Y, Sun J, Yan H, Fan Y, Zhang X, Li Z, Liu X. Neoadjuvant chemo-immunotherapy with camrelizumab plus nab-paclitaxel and cisplatin in resectable locally advanced squamous cell carcinoma of the head and neck: a pilot phase II trial. Nat Commun. 2024 Mar 11;15(1):2177. doi: 10.1038/s41467-024-46444-z. PMID 38467604
- [Background] Gatta G, Botta L, Sanchez MJ, Anderson LA, Pierannunzio D, Licitra L; EUROCARE Working Group:. Prognoses and improvement for head and neck cancers diagnosed in Europe in early 2000s: The EUROCARE-5 population-based study. Eur J Cancer. 2015 Oct;51(15):2130-2143. doi: 10.1016/j.ejca.2015.07.043. Epub 2015 Sep 26. PMID 26421817
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338